CLINICAL TRIAL: NCT06775145
Title: Therapeutic Effect of Neuromodulation on Anxiety Disorders by High-Definition Transcranial Electrical Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202312116DINB
Record Dates: First submitted 2025-01-02; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HD-R_cDC+cTBS & sham-L_aDC+iTBS (Experimental)
  Interventions: Device: HD-R_cDC+cTBS & sham-L_aDC+iTBS
- sham-R_cDC+cTBS & HD-L_aDC+iTBS (Experimental)
  Interventions: Device: sham-R_cDC+cTBS & HD-L_aDC+iTBS
- HD-R_cDC+cTBS & HD-L_aDC+iTBS (Experimental)
  Interventions: Device: HD-R_cDC+cTBS & HD-L_aDC+iTBS
- sham-R_cDC+cTBS & sham-L_aDC+iTBS (Sham Comparator)
  Interventions: Device: sham-R_cDC+cTBS & sham-L_aDC+iTBS

INTERVENTIONS:
Device: HD-R_cDC+cTBS & sham-L_aDC+iTBS — HD-tES inhibitory waveform (cDC+cTBS) applied to the right dorsolateral prefrontal cortex (DLPFC) for 10 minutes, followed by sham excitatory waveform (aDC+iTBS) stimulation applied to the left DLPFC for 10 minutes.
  Arms: HD-R_cDC+cTBS & sham-L_aDC+iTBS
Device: sham-R_cDC+cTBS & HD-L_aDC+iTBS — Sham inhibitory waveform (cDC+cTBS) stimulation applied to the right DLPFC for 10 minutes, followed by HD-tES excitatory waveform (aDC+iTBS) applied to the left DLPFC for 10 minutes.
  Arms: sham-R_cDC+cTBS & HD-L_aDC+iTBS
Device: HD-R_cDC+cTBS & HD-L_aDC+iTBS — HD-tES inhibitory waveform (cDC+cTBS) applied to the right DLPFC for 10 minutes, followed by HD-tES excitatory waveform (aDC+iTBS) applied to the left DLPFC for 10 minutes.
  Arms: HD-R_cDC+cTBS & HD-L_aDC+iTBS
Device: sham-R_cDC+cTBS & sham-L_aDC+iTBS — Sham inhibitory waveform (cDC+cTBS) stimulation applied to the right DLPFC for 10 minutes, followed by sham excitatory waveform (aDC+iTBS) stimulation applied to the left DLPFC for 10 minutes.
  Arms: sham-R_cDC+cTBS & sham-L_aDC+iTBS

SUMMARY:
High-definition transcranial electrical stimulation (HD-tES) is a non-invasive brain neuromodulation technique that applies a small electrical current to the scalp to alter neural excitability and stimulate localized brain activation. Previous clinical trials have explored the use of HD-tES for treating mental health conditions such as depression, anxiety, obsessive-compulsive disorder, and post-traumatic stress disorder. This trial aims to investigate the efficacy and safety of HD-tES in ameliorating anxiety symptoms among patients with generalized anxiety disorder (GAD), thereby validating its potential as a treatment for anxiety disorders.

Participants will be randomly assigned to one of four HD-tES treatment groups: (1) HD-tES inhibitory waveform (cDC+cTBS) applied to the right dorsolateral prefrontal cortex (DLPFC) for 10 minutes, followed by sham excitatory waveform (aDC+iTBS) stimulation applied to the left DLPFC for 10 minutes. (2) Sham inhibitory waveform (cDC+cTBS) stimulation applied to the right DLPFC for 10 minutes, followed by HD-tES excitatory waveform (aDC+iTBS) applied to the left DLPFC for 10 minutes. (3) HD-tES inhibitory waveform (cDC+cTBS) applied to the right DLPFC for 10 minutes, followed by HD-tES excitatory waveform (aDC+iTBS) applied to the left DLPFC for 10 minutes. (4) Sham inhibitory waveform (cDC+cTBS) stimulation applied to the right DLPFC for 10 minutes, followed by sham excitatory waveform (aDC+iTBS) stimulation applied to the left DLPFC for 10 minutes. Regardless of the group assignment, participants will undergo treatment sessions over a 2-week period, with five sessions per week and no more than one session per day. Each session lasts approximately 20 minutes. Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Diagnosed with Generalized Anxiety Disorder (GAD) by a psychiatrist according to DSM-5 criteria.
* Hamilton Anxiety Rating Scale (HAM-A) score ≥ 14.
* Hamilton Depression Rating Scale (HAM-D; 17-item version) score ≤ 17.
* Has been consistently receiving psychological counseling and/or medication with stable types and dosages for at least 6 weeks prior to enrollment; or is deemed unsuitable for medication and/or psychological counseling; or refuses medication and/or psychological counseling.

Exclusion Criteria:

* Received rTMS or any other form of non-invasive brain stimulation techniques within 2 weeks prior to the study and during the study period.
* Presence of severe neurological disorders (e.g., stroke, brain tumor, epilepsy, organic brain diseases) or psychiatric disorders (e.g., schizophrenia and other psychotic disorders, bipolar disorder, obsessive-compulsive disorder, other types of anxiety disorders, substance abuse).
* Severe or unstable physiological conditions that may affect the autonomic or central nervous system (e.g., acute gastrointestinal diseases, cardiovascular diseases, thyroid disorders).
* History of cardiac arrhythmia.
* Presence of implanted medical electronic devices (e.g., pacemakers).
* Presence of metallic implants in the head or neck region.
* Open wounds on the scalp at the site of electrode contact.
* History of head surgery or significant head trauma that, based on physician evaluation, makes the individual unsuitable for inclusion.
* Individuals with significant suicide risk (HAM-D Item 3 score on suicidal risk ≥ 3).
* Presence of immune disorders (e.g., systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, inflammatory bowel diseases).
* Individuals with abnormal or heightened sensitivity to electrical stimulation, making them unable to tolerate it.
* Pregnancy (for female participants: must be postmenopausal or surgically sterilized. Females of childbearing potential must have a negative pregnancy test. Female participants capable of becoming pregnant and their male partners with female partners capable of becoming pregnant must agree to use effective contraception during the trial and for 4 months after the last study intervention, such as oral contraceptives, dual barrier methods, or intrauterine devices, or agree to abstain from sexual activity during this period. Non-childbearing females are defined as those who have undergone bilateral oophorectomy or are postmenopausal).
* Taking medications that lower the seizure threshold.
* Alcohol or substance abuse.
* Convexity skull defects or elevated intracranial pressure.
* Breastfeeding women.
* Other conditions deemed unsuitable for transcranial electrical stimulation based on physician evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in severity of anxious symptoms as assessed by Hamilton Anxiety Rating Scale (HAM-A) and after intervention | Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.
Change in state and trait anxiety as assessed by State-Trait Anxiety Inventory (STAI) after intervention | Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.

SECONDARY OUTCOMES:
Change in severity of depressive symptoms as assessed by Hamilton Depression Scale (HAM-D) after intervention | Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.
Change in sleep quality as assessed by Pittsburgh Sleep Quality Index (PSQI) after intervention | Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.
Self-rated anxiety level as assessed by Visual Analog Scale (VAS) | Within 3 minute after each intervention session (a total of 10 sessions, 5 sessions/week, lasting 2 weeks)
Heart Rate Variability (HRV) as assessed by NeXus-10MK Ⅱ | Within 10 minutes after each intervention session (a total of 10 sessions, 5 sessions/week, lasting 2 weeks)
Side effects as assessed by Side Effects Questionnaire | Within 10 minutes after each intervention session (a total of 10 sessions, 5 sessions/week, lasting 2 weeks)

OTHER OUTCOMES:
Change in working memory ability as assessed by N-back task after intervention | Assessments will be conducted before the treatment, weekly during the treatment period (at the end of the first and second weeks), and a follow-up evaluation will be performed one week after the conclusion of the treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nitsche MA, Doemkes S, Karakose T, Antal A, Liebetanz D, Lang N, Tergau F, Paulus W. Shaping the effects of transcranial direct current stimulation of the human motor cortex. J Neurophysiol. 2007 Apr;97(4):3109-17. doi: 10.1152/jn.01312.2006. Epub 2007 Jan 24. PMID 17251360
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Williams JA, Imamura M, Fregni F. Updates on the use of non-invasive brain stimulation in physical and rehabilitation medicine. J Rehabil Med. 2009 Apr;41(5):305-11. doi: 10.2340/16501977-0356. PMID 19363560
- [Background] Reed T, Cohen Kadosh R. Transcranial electrical stimulation (tES) mechanisms and its effects on cortical excitability and connectivity. J Inherit Metab Dis. 2018 Jul 13;41(6):1123-30. doi: 10.1007/s10545-018-0181-4. Online ahead of print. PMID 30006770
- [Background] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Background] Polania R, Nitsche MA, Ruff CC. Studying and modifying brain function with non-invasive brain stimulation. Nat Neurosci. 2018 Feb;21(2):174-187. doi: 10.1038/s41593-017-0054-4. Epub 2018 Jan 8. PMID 29311747
- [Background] Hummel FC, Voller B, Celnik P, Floel A, Giraux P, Gerloff C, Cohen LG. Effects of brain polarization on reaction times and pinch force in chronic stroke. BMC Neurosci. 2006 Nov 3;7:73. doi: 10.1186/1471-2202-7-73. PMID 17083730
- [Background] Guleyupoglu B, Febles N, Minhas P, Hahn C, Bikson M. Reduced discomfort during high-definition transcutaneous stimulation using 6% benzocaine. Front Neuroeng. 2014 Jul 11;7:28. doi: 10.3389/fneng.2014.00028. eCollection 2014. PMID 25071548
- [Background] Turski CA, Kessler-Jones A, Chow C, Hermann B, Hsu D, Jones J, Seeger SK, Chappell R, Boly M, Ikonomidou C. Extended Multiple-Field High-Definition transcranial direct current stimulation (HD-tDCS) is well tolerated and safe in healthy adults. Restor Neurol Neurosci. 2017;35(6):631-642. doi: 10.3233/RNN-170757. PMID 29172010
- [Background] Kuo HI, Bikson M, Datta A, Minhas P, Paulus W, Kuo MF, Nitsche MA. Comparing cortical plasticity induced by conventional and high-definition 4 x 1 ring tDCS: a neurophysiological study. Brain Stimul. 2013 Jul;6(4):644-8. doi: 10.1016/j.brs.2012.09.010. Epub 2012 Oct 13. PMID 23149292
- [Background] Cox J, Thakur B, Alvarado L, Shokar N, Thompson PM, Dwivedi AK. Repetitive transcranial magnetic stimulation for generalized anxiety and panic disorders: A systematic review and meta-analysis. Ann Clin Psychiatry. 2022 May;34(2):e2-e24. doi: 10.12788/acp.0050. PMID 35550035
- [Background] de Lima AL, Braga FMA, da Costa RMM, Gomes EP, Brunoni AR, Pegado R. Transcranial direct current stimulation for the treatment of generalized anxiety disorder: A randomized clinical trial. J Affect Disord. 2019 Dec 1;259:31-37. doi: 10.1016/j.jad.2019.08.020. Epub 2019 Aug 15. PMID 31437698
- [Background] Diefenbach GJ, Bragdon LB, Zertuche L, Hyatt CJ, Hallion LS, Tolin DF, Goethe JW, Assaf M. Repetitive transcranial magnetic stimulation for generalised anxiety disorder: a pilot randomised, double-blind, sham-controlled trial. Br J Psychiatry. 2016 Sep;209(3):222-8. doi: 10.1192/bjp.bp.115.168203. Epub 2016 May 19. PMID 27198484
- [Background] Dilkov D, Hawken ER, Kaludiev E, Milev R. Repetitive transcranial magnetic stimulation of the right dorsal lateral prefrontal cortex in the treatment of generalized anxiety disorder: A randomized, double-blind sham controlled clinical trial. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Aug 1;78:61-65. doi: 10.1016/j.pnpbp.2017.05.018. Epub 2017 May 19. PMID 28533148
- [Background] Huang Z, Li Y, Bianchi MT, Zhan S, Jiang F, Li N, Ding Y, Hou Y, Wang L, Ouyang Q, Wang Y. Repetitive transcranial magnetic stimulation of the right parietal cortex for comorbid generalized anxiety disorder and insomnia: A randomized, double-blind, sham-controlled pilot study. Brain Stimul. 2018 Sep-Oct;11(5):1103-1109. doi: 10.1016/j.brs.2018.05.016. Epub 2018 May 29. PMID 29871798
- [Background] Labree B, Hoare DJ, Gascoyne LE, Scutt P, Del Giovane C, Sereda M. Determining the Effects of Transcranial Direct Current Stimulation on Tinnitus, Depression, and Anxiety: A Systematic Review. Brain Sci. 2022 Apr 8;12(4):484. doi: 10.3390/brainsci12040484. PMID 35448015
- [Background] Nasiri F, Mashhadi A, Bigdeli I, Chamanabad AG, Ellard KK. Augmenting the unified protocol for transdiagnostic treatment of emotional disorders with transcranial direct current stimulation in individuals with generalized anxiety disorder and comorbid depression: A randomized controlled trial. J Affect Disord. 2020 Feb 1;262:405-413. doi: 10.1016/j.jad.2019.11.064. Epub 2019 Nov 11. PMID 31740106
- [Background] Sadeghi Movahed, F., et al., Effectiveness of Transcranial Direct Current Stimulation on Worry, Anxiety, and Depression in Generalized Anxiety Disorder: A Randomized, Single-Blind Pharmacotherapy and Sham- Controlled Clinical Trial. Iran J Psychiatry Behav Sci, 2018. 12(2): p. e11071.
- [Background] Vergallito A, Gallucci A, Pisoni A, Punzi M, Caselli G, Ruggiero GM, Sassaroli S, Romero Lauro LJ. Effectiveness of noninvasive brain stimulation in the treatment of anxiety disorders: a meta-analysis of sham or behaviour-controlled studies. J Psychiatry Neurosci. 2021 Nov 9;46(6):E592-E614. doi: 10.1503/jpn.210050. Print 2021 Nov-Dec. PMID 34753789
- [Background] McPhee ME, Graven-Nielsen T. Medial Prefrontal High-Definition Transcranial Direct Current Stimulation to Improve Pain Modulation in Chronic Low Back Pain: A Pilot Randomized Double-blinded Placebo-Controlled Crossover Trial. J Pain. 2021 Aug;22(8):952-967. doi: 10.1016/j.jpain.2021.02.012. Epub 2021 Mar 4. PMID 33676009
- [Background] Santana K, Franca E, Sato J, Silva A, Queiroz M, de Farias J, Rodrigues D, Souza I, Ribeiro V, Caparelli-Daquer E, Teixeira AL, Charvet L, Datta A, Bikson M, Andrade S. Non-invasive brain stimulation for fatigue in post-acute sequelae of SARS-CoV-2 (PASC). Brain Stimul. 2023 Jan-Feb;16(1):100-107. doi: 10.1016/j.brs.2023.01.1672. Epub 2023 Jan 21. PMID 36693536
- [Background] Li YT, Chen SC, Yang LY, Hsieh TH, Peng CW. Designing and Implementing a Novel Transcranial Electrostimulation System for Neuroplastic Applications: A Preliminary Study. IEEE Trans Neural Syst Rehabil Eng. 2019 May;27(5):805-813. doi: 10.1109/TNSRE.2019.2908674. Epub 2019 Apr 2. PMID 30951469
- [Background] Huang YJ, Wang SM, Chen C, Chen CA, Wu CW, Chen JJ, Peng CW, Lin CW, Huang SW, Chen SC. High-Definition Transcranial Direct Current with Electrical Theta Burst on Post-Stroke Motor Rehabilitation: A Pilot Randomized Controlled Trial. Neurorehabil Neural Repair. 2022 Sep;36(9):645-654. doi: 10.1177/15459683221121751. Epub 2022 Sep 1. PMID 36047662
- [Background] Wang SS, Huang YJ, Chen JJ, Wu CW, Chen CA, Lin CW, Nguyen VT, Peng CW. Designing and pilot testing a novel high-definition transcranial burst electrostimulation device for neurorehabilitation. J Neural Eng. 2021 Sep 17;18(5). doi: 10.1088/1741-2552/ac23be. PMID 34479230
- [Background] Stagg CJ, Bachtiar V, O'Shea J, Allman C, Bosnell RA, Kischka U, Matthews PM, Johansen-Berg H. Cortical activation changes underlying stimulation-induced behavioural gains in chronic stroke. Brain. 2012 Jan;135(Pt 1):276-84. doi: 10.1093/brain/awr313. Epub 2011 Dec 6. PMID 22155982
- [Background] Bologna M, Paparella G, Fabbrini A, Leodori G, Rocchi L, Hallett M, Berardelli A. Effects of cerebellar theta-burst stimulation on arm and neck movement kinematics in patients with focal dystonia. Clin Neurophysiol. 2016 Nov;127(11):3472-3479. doi: 10.1016/j.clinph.2016.09.008. Epub 2016 Sep 15. PMID 27721106
- [Background] Cao L, Fu W, Zhang Y, Huo S, Du J, Zhu L, Song W. Intermittent theta burst stimulation modulates resting-state functional connectivity in the attention network and promotes behavioral recovery in patients with visual spatial neglect. Neuroreport. 2016 Dec 7;27(17):1261-1265. doi: 10.1097/WNR.0000000000000689. PMID 27748671
- [Background] Vanbellingen T, Wapp M, Stegmayer K, Bertschi M, Abela E, Kubel S, Nyffeler T, Muri R, Walther S, Nef T, Hallett M, Bohlhalter S. Theta burst stimulation over premotor cortex in Parkinson's disease: an explorative study on manual dexterity. J Neural Transm (Vienna). 2016 Dec;123(12):1387-1393. doi: 10.1007/s00702-016-1614-6. Epub 2016 Sep 12. PMID 27619658
- [Background] Wu CW, Chiu WT, Hsieh TH, Hsieh CH, Chen JJ. Modulation of motor excitability by cortical optogenetic theta burst stimulation. PLoS One. 2018 Aug 30;13(8):e0203333. doi: 10.1371/journal.pone.0203333. eCollection 2018. PMID 30161250
- [Background] Hsieh, T.-H., et al., Novel Use of Theta Burst Cortical Electrical Stimulation for Modulating Motor Plasticity in Rats. Journal of Medical and Biological Engineering, 2015. 35(1): p. 62-68.
- [Background] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Background] Nitsche MA, Schauenburg A, Lang N, Liebetanz D, Exner C, Paulus W, Tergau F. Facilitation of implicit motor learning by weak transcranial direct current stimulation of the primary motor cortex in the human. J Cogn Neurosci. 2003 May 15;15(4):619-26. doi: 10.1162/089892903321662994. PMID 12803972
- [Background] Datta A, Bansal V, Diaz J, Patel J, Reato D, Bikson M. Gyri-precise head model of transcranial direct current stimulation: improved spatial focality using a ring electrode versus conventional rectangular pad. Brain Stimul. 2009 Oct;2(4):201-7, 207.e1. doi: 10.1016/j.brs.2009.03.005. PMID 20648973
- [Background] Albein-Urios N, Chase H, Clark L, Kirkovski M, Davies C, Enticott PG. Increased perseverative errors following high-definition transcranial direct current stimulation over the ventrolateral cortex during probabilistic reversal learning. Brain Stimul. 2019 Jul-Aug;12(4):959-966. doi: 10.1016/j.brs.2019.02.013. Epub 2019 Feb 21. PMID 30833215
- [Background] Chua EF, Ahmed R, Garcia SM. Effects of HD-tDCS on memory and metamemory for general knowledge questions that vary by difficulty. Brain Stimul. 2017 Mar-Apr;10(2):231-241. doi: 10.1016/j.brs.2016.10.013. Epub 2016 Nov 1. PMID 27876306
- [Background] Doppelmayr M, Pixa NH, Steinberg F. Cerebellar, but not Motor or Parietal, High-Density Anodal Transcranial Direct Current Stimulation Facilitates Motor Adaptation. J Int Neuropsychol Soc. 2016 Oct;22(9):928-936. doi: 10.1017/S1355617716000345. Epub 2016 May 6. PMID 27152869
- [Background] Gozenman F, Berryhill ME. Working memory capacity differentially influences responses to tDCS and HD-tDCS in a retro-cue task. Neurosci Lett. 2016 Aug 26;629:105-109. doi: 10.1016/j.neulet.2016.06.056. Epub 2016 Jun 28. PMID 27369325
- [Background] Hogeveen J, Grafman J, Aboseria M, David A, Bikson M, Hauner KK. Effects of High-Definition and Conventional tDCS on Response Inhibition. Brain Stimul. 2016 Sep-Oct;9(5):720-729. doi: 10.1016/j.brs.2016.04.015. Epub 2016 Apr 22. PMID 27198577
- [Background] Muthalib M, Besson P, Rothwell J, Perrey S. Focal Hemodynamic Responses in the Stimulated Hemisphere During High-Definition Transcranial Direct Current Stimulation. Neuromodulation. 2018 Jun;21(4):348-354. doi: 10.1111/ner.12632. Epub 2017 Jul 17. PMID 28714545
- [Background] Muthalib M, Besson P, Rothwell J, Ward T, Perrey S. Effects of Anodal High-Definition Transcranial Direct Current Stimulation on Bilateral Sensorimotor Cortex Activation During Sequential Finger Movements: An fNIRS Study. Adv Exp Med Biol. 2016;876:351-359. doi: 10.1007/978-1-4939-3023-4_44. PMID 26782232
- [Background] Nikolin S, Lauf S, Loo CK, Martin D. Effects of High-Definition Transcranial Direct Current Stimulation (HD-tDCS) of the Intraparietal Sulcus and Dorsolateral Prefrontal Cortex on Working Memory and Divided Attention. Front Integr Neurosci. 2019 Jan 8;12:64. doi: 10.3389/fnint.2018.00064. eCollection 2018. PMID 30670954
- [Background] Nikolin S, Loo CK, Bai S, Dokos S, Martin DM. Focalised stimulation using high definition transcranial direct current stimulation (HD-tDCS) to investigate declarative verbal learning and memory functioning. Neuroimage. 2015 Aug 15;117:11-9. doi: 10.1016/j.neuroimage.2015.05.019. Epub 2015 May 15. PMID 25987365
- [Background] Pixa NH, Steinberg F, Doppelmayr M. High-definition transcranial direct current stimulation to both primary motor cortices improves unimanual and bimanual dexterity. Neurosci Lett. 2017 Mar 16;643:84-88. doi: 10.1016/j.neulet.2017.02.033. Epub 2017 Feb 14. PMID 28229937
- [Background] Reckow J, Rahman-Filipiak A, Garcia S, Schlaefflin S, Calhoun O, DaSilva AF, Bikson M, Hampstead BM. Tolerability and blinding of 4x1 high-definition transcranial direct current stimulation (HD-tDCS) at two and three milliamps. Brain Stimul. 2018 Sep-Oct;11(5):991-997. doi: 10.1016/j.brs.2018.04.022. Epub 2018 May 4. PMID 29784589
- [Background] Heimrath K, Breitling C, Krauel K, Heinze HJ, Zaehle T. Modulation of pre-attentive spectro-temporal feature processing in the human auditory system by HD-tDCS. Eur J Neurosci. 2015 Jun;41(12):1580-6. doi: 10.1111/ejn.12908. Epub 2015 May 8. PMID 25847301
- [Background] Gbadeyan O, McMahon K, Steinhauser M, Meinzer M. Stimulation of Dorsolateral Prefrontal Cortex Enhances Adaptive Cognitive Control: A High-Definition Transcranial Direct Current Stimulation Study. J Neurosci. 2016 Dec 14;36(50):12530-12536. doi: 10.1523/JNEUROSCI.2450-16.2016. PMID 27974612
- [Background] Fiori V, Nitsche MA, Cucuzza G, Caltagirone C, Marangolo P. High-Definition Transcranial Direct Current Stimulation Improves Verb Recovery in Aphasic Patients Depending on Current Intensity. Neuroscience. 2019 May 15;406:159-166. doi: 10.1016/j.neuroscience.2019.03.010. Epub 2019 Mar 12. PMID 30876982
- [Background] Caparelli-Daquer EM, Zimmermann TJ, Mooshagian E, Parra LC, Rice JK, Datta A, Bikson M, Wassermann EM. A pilot study on effects of 4x1 high-definition tDCS on motor cortex excitability. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:735-8. doi: 10.1109/EMBC.2012.6346036. PMID 23365997
- [Background] Kessler SK, Turkeltaub PE, Benson JG, Hamilton RH. Differences in the experience of active and sham transcranial direct current stimulation. Brain Stimul. 2012 Apr;5(2):155-62. doi: 10.1016/j.brs.2011.02.007. Epub 2011 Mar 27. PMID 22037128
- [Background] Villamar MF, Wivatvongvana P, Patumanond J, Bikson M, Truong DQ, Datta A, Fregni F. Focal modulation of the primary motor cortex in fibromyalgia using 4x1-ring high-definition transcranial direct current stimulation (HD-tDCS): immediate and delayed analgesic effects of cathodal and anodal stimulation. J Pain. 2013 Apr;14(4):371-83. doi: 10.1016/j.jpain.2012.12.007. Epub 2013 Feb 14. PMID 23415877
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Bulteau S, Sebille V, Fayet G, Thomas-Ollivier V, Deschamps T, Bonnin-Rivalland A, Laforgue E, Pichot A, Valriviere P, Auffray-Calvier E, Fortin J, Pereon Y, Vanelle JM, Sauvaget A. Efficacy of intermittent Theta Burst Stimulation (iTBS) and 10-Hz high-frequency repetitive transcranial magnetic stimulation (rTMS) in treatment-resistant unipolar depression: study protocol for a randomised controlled trial. Trials. 2017 Jan 13;18(1):17. doi: 10.1186/s13063-016-1764-8. PMID 28086851
- [Background] Demirtas-Tatlidede A, Vahabzadeh-Hagh AM, Bernabeu M, Tormos JM, Pascual-Leone A. Noninvasive brain stimulation in traumatic brain injury. J Head Trauma Rehabil. 2012 Jul-Aug;27(4):274-92. doi: 10.1097/HTR.0b013e318217df55. PMID 21691215
- [Background] Galhardoni R, Correia GS, Araujo H, Yeng LT, Fernandes DT, Kaziyama HH, Marcolin MA, Bouhassira D, Teixeira MJ, de Andrade DC. Repetitive transcranial magnetic stimulation in chronic pain: a review of the literature. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S156-72. doi: 10.1016/j.apmr.2014.11.010. Epub 2014 Nov 28. PMID 25437106
- [Background] Miniussi C, Rossini PM. Transcranial magnetic stimulation in cognitive rehabilitation. Neuropsychol Rehabil. 2011 Oct;21(5):579-601. doi: 10.1080/09602011.2011.562689. Epub 2011 Jun 24. PMID 21462081
- [Background] Chen YJ, Huang YZ, Chen CY, Chen CL, Chen HC, Wu CY, Lin KC, Chang TL. Intermittent theta burst stimulation enhances upper limb motor function in patients with chronic stroke: a pilot randomized controlled trial. BMC Neurol. 2019 Apr 25;19(1):69. doi: 10.1186/s12883-019-1302-x. PMID 31023258
- [Background] Hsu WY, Cheng CH, Liao KK, Lee IH, Lin YY. Effects of repetitive transcranial magnetic stimulation on motor functions in patients with stroke: a meta-analysis. Stroke. 2012 Jul;43(7):1849-57. doi: 10.1161/STROKEAHA.111.649756. Epub 2012 Jun 19. PMID 22713491
- [Background] Shin J, Yang E, Cho K, Barcenas CL, Kim WJ, Min Y, Paik NJ. Clinical application of repetitive transcranial magnetic stimulation in stroke rehabilitation. Neural Regen Res. 2012 Mar 15;7(8):627-34. doi: 10.3969/j.issn.1673-5374.2012.08.011. PMID 25745455
- [Background] Jaberzadeh S, Bastani A, Zoghi M. Anodal transcranial pulsed current stimulation: A novel technique to enhance corticospinal excitability. Clin Neurophysiol. 2014 Feb;125(2):344-51. doi: 10.1016/j.clinph.2013.08.025. Epub 2013 Sep 26. PMID 24074626
- [Background] Morales-Quezada L, Cosmo C, Carvalho S, Leite J, Castillo-Saavedra L, Rozisky JR, Fregni F. Cognitive effects and autonomic responses to transcranial pulsed current stimulation. Exp Brain Res. 2015 Mar;233(3):701-9. doi: 10.1007/s00221-014-4147-y. Epub 2014 Dec 6. PMID 25479736
- [Background] Kunz P, Antal A, Hewitt M, Neef A, Opitz A, Paulus W. 5 kHz Transcranial Alternating Current Stimulation: Lack of Cortical Excitability Changes When Grouped in a Theta Burst Pattern. Front Hum Neurosci. 2017 Jan 10;10:683. doi: 10.3389/fnhum.2016.00683. eCollection 2016. PMID 28119589
- [Background] Miller JP, Sweet JA, Bailey CM, Munyon CN, Luders HO, Fastenau PS. Visual-spatial memory may be enhanced with theta burst deep brain stimulation of the fornix: a preliminary investigation with four cases. Brain. 2015 Jul;138(Pt 7):1833-42. doi: 10.1093/brain/awv095. Epub 2015 Apr 21. PMID 26106097
- [Background] Brunye TT, Patterson JE, Wooten T, Hussey EK. A Critical Review of Cranial Electrotherapy Stimulation for Neuromodulation in Clinical and Non-clinical Samples. Front Hum Neurosci. 2021 Feb 1;15:625321. doi: 10.3389/fnhum.2021.625321. eCollection 2021. PMID 33597854